CLINICAL TRIAL: NCT02420171
Title: Adding Insulin to IVF Culture Media Significantly Improve Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banon IVF Center Assiut, Egypt (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Laboratory Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Ibnsina IVF center Sohag
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Infertility
Keywords: In Vitro; embryo quality; Intracytoplasmic sperm injection
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- In Vitro culture media with insulin (Active Comparator): We will add insulin to the single step culture media to monitor the embryogenesis
  Interventions: Other: Adding insulin to In Vitro culture media
- In Vitro culture media without insulin m (No Intervention): The embryos will be cultured in the media without insulin and compare this arm as the control arm with the interventional one.

INTERVENTIONS:
Other: Adding insulin to In Vitro culture media — We will add insulin for in vitro culture of human embryos
  Arms: In Vitro culture media with insulin

SUMMARY:
Add insulin to a single step culture media for IVF embryo culture from day 0 to day 5/6 of In Vitro culture and detect the the effect upon embryo quality and implantation potential.

DETAILED DESCRIPTION:
The IVF culture media design and upgrade underwent many ideas during the last 3 decades, we suppose that adding insulin as a hormon and growth factor might improve embryo development in vitro so we decide to design a trial to compare the embryogenesis by sibling Oocytes of the same patient between to arm of the same culture media and yhe same culture condition but with one arm with insulin and the other is traditional one and closely monitor the outcome within the 2 arms abd record the results

ELIGIBILITY:
Inclusion Criteria:

* normal responder
* PCOS
* Tubal factor infertility
* mild asthenozoospermia

Exclusion Criteria:

* patient over 40

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
clinical Pregnancy rate ( % ) | 6 months

SECONDARY OUTCOMES:
Blastocyst rate ( % ) | 6 months
Blastocyst quality rate ( % ) | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Banon IVF Center, Asyut
  - Ibnsina IVF center, Sohag